CLINICAL TRIAL: NCT02557464
Title: Identification of Early Semantic Markers of Alzheimer's Disease by Using Eye Tracking in Reading Neutral and Predictable Sentences
Brief Title: Identification of Early Markers of Alzheimer's Disease by Using Eye Tracking in Reading.
Acronym: ADAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-AOI-04
Record Dates: First submitted 2015-09-10; First posted 2015-09-23 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer's Disease
Keywords: semantic memory; eye movements; reading
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alzheimer's disease group (Experimental): 24 patients with an Alzheimer's disease or related disorders
  Interventions: Behavioral: An eye tracking experiment; Behavioral: A neuropsychological evaluation
- control group (Active Comparator): 24 age matched controls participants
  Interventions: Behavioral: An eye tracking experiment; Behavioral: A neuropsychological evaluation

INTERVENTIONS:
Behavioral: An eye tracking experiment — Neuropsychological assessments and eye tracking during reading will be practice twice with an interval of 6 months
Behavioral: A neuropsychological evaluation — Neuropsychological assessments and eye tracking during reading will be practice twice with an interval of 6 months

SUMMARY:
The objective of this study is to identify early and accurate semantics markers of Alzheimer's disease (AD) by using two types of methods. First, the investigator will evaluate semantic processing of patients with AD or related disorders which will be compared to age matched controls by taking neuropsychological tests. Then, the investigator will analyze the effect of contextual word predictability on eye movements in reading sentences with the help of the same participants by using an eye tracker. Both of these methods will be used twice with a time interval of 6 months.

DETAILED DESCRIPTION:
Scientific background:

Identifying Alzheimer's disease (AD) as early as possible should enable to propose a re-education platform that would fit the early stage of neuronal loss in this pathology. Neuropsychological evaluations are currently one of the main tools for the early screening of AD. Among the tests proposed during those evaluations, the investigator find the Isaacs Set Test which evaluates the early degradation of semantic memory. Whereas eyes movement behavior during reading is sensitive to semantics factors and allows collecting accurate measurements (as precisely as one millisecond), no study has yet used this technique to precisely identify the precocious semantics troubles of AD.

Goal:

The objective of this study is to identify early and accurate markers of AD by associating semantic neuropsychological assessments and eye tracking during sentences reading.

Method:

The study will include 24 patients with AD or related disorders (Mini Mental State Examination between 20 and 27 ) and 24 age matched controls participants. The experiment will be divided in two steps. First, patients will take a standard neuropsychological evaluation. A specific semantic analysis will be performed on each participant using, for example, the Isaacs Set Test or the Weschler Similarities. The second step will ask the participants to read sentences while an eye tracker (the Eye Link 1000 remote) will record their eyes movements. In order to manipulate semantics factors, each sentence will contain a target word, either predictable or not. The experiment will last one hour and a half. Neuropsychological assessments and eye tracking will be done twice with a time interval of 6 months. The two times will be called T1 and T2 and are required to estimate whether eye tracking is a better predictor of AD than neuropsychological tests or not.

Evaluation criteria:

The eye tracking technique enables to record different sorts of measures. More specifically, the investigator will evaluate gaze duration on the target word. Moreover, neuropsychological tests scores will be collected. It will be, for example, the number of good answers.

Hypothesis and expected results:

First, the investigator expect that the predictability effect on eye movements would be less pronounced for patients with AD or related disorders than for the control group. This effect would be even more diminished at T2. It could be explained by a progressive degradation of the semantic memory of patients. Then, and for the same reasons, the investigator expect that the scores collected from the neuropsychological tests would be pathological for patient suffering from AD or related disorders. The test scores would be even more in deficit at T2. Finally, the investigator predict a correlation between neuropsychological tests data and eye movements data. With an extrapolation, and because eye movements recording allow us to obtain more accurate information about the quality of semantic processes, the investigator formulate the hypothesis that this technique will help to predict earlier AD.

ELIGIBILITY:
Inclusion Criteria:

Pour le bras A :

Inclusion criteria

* Mother tongue french participants
* Participants with a level of education = or > to Junior Secondary School Diploma
* Participants with a normal or corrected vision
* Participants with good score at the neuro visual assessments (> or = to 15 at the "detection test" ; > or = to 16 at the "degraded letters" test
* Participants suffering from Alzheimer's or related disorders disease (ICD-10 criteria)
* Participants with an MMSE's score between 20 and 27
* Participants must sign the informed consent
* Participants must be affiliated to the social insurance. Non-inclusion criteria
* Impossibility to realize the experiment because of a blurred vision
* History of neurological or psychiatric disease, of alcoholism and of brain injury
* Participants under trusteeship, guardianship or placed under judicial protection
* Persons deprived of their liberty

Pour le bras B :

Inclusion criteria

* Mother tongue french participants
* Participants with a level of education = or > to Junior Secondary School Diploma
* Participants with a normal or corrected vision
* Participants with no global cognitive impairment with a MMSE's score > or = to 28 and with no difficulty to repeat and recall the 3 words
* Participants with good score at the neuro visual assessments (> or = to 15 at the "detection test" ; > or = to 16 at the "degraded letters" test
* Participants must sign the informed consent
* Participants must be affiliated to the social insurance. Non-inclusion criteria
* Impossibility to realize the experiment because of a blurred vision
* Prescription of psychotropic medication during the week preceding the experiment
* History of neurological or psychiatric disease, of alcoholism and of brain injury
* Evidence of cognitive decline
* Decline in the day-to-day operations
* Participants under trusteeship, guardianship or placed under judicial protection
* Persons deprived of their liberty

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Eye tracking | at six months
  Eye tracking (More specifically, the investigator will evaluate gaze duration on target words included in sentences while participant's eye movements will be recorded with the Eye link 1000 remote. Gaze duration is the sum of all fixations on a word prior to moving to another word)

SECONDARY OUTCOMES:
The probability that the eyes skip the target word | at six months
  The Visual Object and Space Perception Battery ( for the "degraded letters" test scores range from 0 to 20 and a score below 16 is considered as pathological; for the "test of detection" scores range from 0 to 20 and a score below 15 is considered as pathological). This test assesses neurovisual capacity
the initial landing position of the eye in the target word (in letters) | at six months
  An eye tracking experiment while participants read sentences on a computer screen
the percentage of refixation done on the target word | at six months
the first fixation duration in the target word | at six months
  (i.e. the duration of the first fixation on the target word, provided that the word wasn't skipped
the single fixation duration | at six months
  the fixation of the target word when only one fixation is made on that word
the percentage of regressive saccade on the target word and the total viewing time | at six months
Neuropsychological tests scores | at six months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claude Pompidou, Nice, France